CLINICAL TRIAL: NCT05399264
Title: Efficacy of Auditory Training and Combined Auditory-working-memory Training in Improving Communication and Cognition in Older Adults With Untreated Mild-to-moderate Sensorineural Hearing Impairment
Brief Title: Efficacy of Auditory Training and Combined Auditory-working-memory Training in Improving Communication in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-2022-0134
Record Dates: First submitted 2022-05-11; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hearing Loss
Keywords: Auditory training; Working memory; Speech perception; Older adults; Hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auditory-working memory training group (Experimental): The auditory-working memory training (AT-WMT) program is home-delivered, non-clinician-administered, and computer-based. That is, training will be self-paced and administered by the participants themselves at home using a computer. A software program has been created to facilitate the administration. Participants will spend one hour per day and five days per week for 4 weeks on training.
  During the training, the following two adaptive tasks will be administered simultaneously: repeating the sentences masked by noise (i.e., AT component) and recalling the first or the final two words of all sentences in a given sentence set (i.e., WMT component).
  Interventions: Behavioral: Auditory-working memory training program
- Adaptive Auditory training group (Active Comparator): The sentences used in the AT program are the same as those in the AT-WMT program. However, only the AT component (i.e., adaptive sentence perception in noise) of the AT-WMT program is required in the AT program. Participants do not need to recall the first or the final two words of the sentences. The same software in the experimental group will be used. Participants will spend one hour per day and five days per week for 4 weeks on training.
  Interventions: Behavioral: Auditory training program
- Mindfulness training group (Placebo Comparator): Participants in this group will participate in a mindfulness training program using newlife.330 (Psychiatric Rehabilitation Association, 2018) which is a Cantonese online platform for self-guided mindfulness training. The time and computer use of the active-control group will match to those of the above two groups.
  Interventions: Behavioral: Mindfulness training program

INTERVENTIONS:
Behavioral: Auditory-working memory training program — The AT-WMT program is comprised of 1,200 daily used sentences either created or selected from newspapers, books, TV programs and magazines by the research assistants. The sentences are political-, cultural-, and religious-neutral sentences. Each of them contains 10 words. Noise was recorded from the upper and lower decks of a bus, in a café, a Chinese restaurant, an MTR (the Mass Transit Railway) carriage, and from a street.
  During the training, the following two adaptive tasks will be administered simultaneously: repeating the sentences masked by noise (i.e., AT component) and recalling the first or the final two words of all sentences in a given sentence set (i.e., WMT component).
  Arms: Auditory-working memory training group
Behavioral: Auditory training program — During the training, an adaptive speech-in-noise perception task will be administered. Specifically, the sentences in a sentence set will be presented binaurally using a headphone at a level the listeners felt is comfortable. The trainees are expected to immediately repeat each noise-masked sentence after hearing it. If they cannot repeat the sentence, then the sound intensity of the noise will be automatically decreased (step size = 2 dB) until the sentence can be correctly repeated. If the sentence can be repeated at the first attempt, then the intensity of the noise will be automatically increased by 2 dB in the next sentence. To provide feedback, the targeted sentence will be replaced by an asterisk and only shown after clicking the sentence.
  Arms: Adaptive Auditory training group
Behavioral: Mindfulness training program — Participants in this group will participate in a mindfulness training program using newlife.330 (Psychiatric Rehabilitation Association, 2018) which is a Cantonese online platform for self-guided mindfulness training.
  Arms: Mindfulness training group

SUMMARY:
Using a randomized controlled trial, we are going to examine whether a training program that incorporates both auditory training and working memory training (AT-WMT) would generate significantly better results in communication and cognition than an auditory training program and a mindfulness training program (active-control). Participants are 120 older adults (40 per group) with untreated mild-to-moderate sensorineural hearing impairment .

DETAILED DESCRIPTION:
There will be three training groups: the Auditory training (AT) group, the Auditory-working memory training (AT-WMT) group, and the control group (mindfulness training). All training programs are home-delivered, non-clinician-administered, and computer-based. That is, training will be self-paced and administered by the participants themselves at home using a computer. A software program (see Figure 2) has been created to facilitate the administration of the AT and AT-WMT. All training groups will spend one hour per day and five days per week for 4 weeks.

Before the training, two baseline test sessions (T1 and T2, a maximum of one week apart) will be used to account for the test-retest effects. The same measurements will be administered again one day (T3) and three months (T4) after completion of the training.

ELIGIBILITY:
Inclusion Criteria:

* Native Cantonese speakers and having been living in Hong Kong for at least 20 years.
* Aged between 55 and 80 years.
* Normal cognitive function, as screened with the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) with a cutoff of 18/19.
* Mild-to-moderate sensorineural HI, in which the four-frequency pure-tone average at 500, 1000, 2000, and 4000 Hz of the better ear is between 26 and 55 dB HL.

Exclusion Criteria:

* Outer or middle ear pathologies.
* Wearing hearing aids or cochlear implants.
* No computers and internet access at home.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The Cantonese version of the Hearing in Noise Test (CHINT) (Changes are being assessed) | One week before the training, one day before the training, one day after the training, three months after the training
  The Cantonese version of the Hearing in Noise Test (CHINT) (Wong & Soli, 2005) will be used to measure sentence perception in noise. The tool contains 12 lists of 20 sentences, and each sentence comprises 10 words. A high inter-list reliability has been previously demonstrated, which suggests that the lists are equivalent and, therefore, consistent results can be obtained using any of the lists (Wong et al., 2005).
The Cantonese version of the reading span test (CRST) (Changes are being assessed) | One week before the training, one day before the training, one day after the training, three months after the training
  The Cantonese version of the reading span test (CRST) with dual task design will be used to measure WM. It was developed based on the German reading span test (Carroll et al., 2015). The reliability and validity of the CRST have been examined to confirm that the CRST is a suitable test for investigating verbal WM (Cheung, 2021).
  The CRST comprises 54 six-word sentences. The sentences are presented in different set sizes (i.e., 3, 4, 5, and 6 sentences) in random order. The participants are expected to read aloud the sentences presented on a computer screen and judge whether the sentence is semantically correct. After reading aloud all sentences in a given sentence set, the participants will be asked to recall the first or last two words of each sentence in the set. The reading span score is based on the second task: the total number of words recalled. Approximately 20 minutes is needed to complete the test.

SECONDARY OUTCOMES:
The CogState Battery (Changes are being assessed) | One week before the training, one day before the training, one day after the training, three months after the training
  Other cognitive functions (executive function, response inhibition, processing speed, and attention) will be examined using the CogState Battery, which is a sensitive computer-based assessment instrument. The test battery has been adapted for Chinese and its reliability and validity have been previously reported (Zhong et al., 2013). The test battery includes the following subtests and uses playing cards, digits, and pictures as stimuli: 1) One Back Test (short-term memory), 2) Groton Maze Learning Test (executive function), 3) Identification Test (Attention), 4) Go/No-Go Test (response inhibition), 5) International Digit Symbol Substitution Test-Symbols (processing speed). Each CogState subtask takes approximately 3-8 minutes. The entire CogState test battery is expected to be completed in 30-45 minutes.
The Speech, Spatial, and Qualities of Hearing scale (SSQHS) (Changes are being assessed) | One week before the training, one day before the training, one day after the training, three months after the training
  The Speech, Spatial, and Qualities of Hearing scale (SSQHS) (Gatehouse & Noble, 2004) will be used to assess abilities and experience of hearing in different listening environments. The SSQHS is assessed using a self-report questionnaire that comprises 49 questions across the following three scales: 1) speech hearing (n = 14) for measuring the ability to recognize speech in a variety of competing contexts; 2) spatial hearing (n = 17) for assessing the ability of the directional, distance, and movement components of spatial hearing; 3) quality of hearing (n = 18) for evaluating the quality of hearing experience, including the clarity and naturalness of different speakers and everyday sounds, and ease of listening. The use of the SSQHS has been validated for Cantonese speakers (Lee, 2015).
Auditory Brainstem Responses to Complex Sounds (Changes are being assessed) | One week before the training, one day before the training, one day after the training, three months after the training
  The stimulus, a 175 milliseconds /ji/ with Cantonese Tone 4 (low falling), will be used for recoding of subcortical neural responses to lexical tone. Stimuli with an interstimulus interval of 80 milliseconds will be presented in alternating polarity at 80 dB SPL and at 10 dB SNR with a six-speaker multi-talker noise through an insert earphone (ER-3, Etymotic Research). This type of noise and SNR were used in previous studies where significant relationships between SIN perception and cABRs were reported (Anderson & Kraus, 2010b; Anderson et al., 2011). Responses will be collected using a vertical electrode montage (ipsilateral earlobe reference, Cz active, and forehead ground) with the SmartEP (Intelligence Hearing Systems). An average of 6,000 sweeps will be made for responses to /ji4/ in quiet and multi-talker babble noise conditions, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yuan, PhD, Principal Investigator — The Education University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong LL, Soli SD. Development of the Cantonese Hearing In Noise Test (CHINT). Ear Hear. 2005 Jun;26(3):276-89. doi: 10.1097/00003446-200506000-00004. PMID 15937409
- [Background] Anderson S, Parbery-Clark A, Yi HG, Kraus N. A neural basis of speech-in-noise perception in older adults. Ear Hear. 2011 Nov-Dec;32(6):750-7. doi: 10.1097/AUD.0b013e31822229d3. PMID 21730859
- [Background] Anderson S, Kraus N. Sensory-cognitive interaction in the neural encoding of speech in noise: a review. J Am Acad Audiol. 2010 Oct;21(9):575-85. doi: 10.3766/jaaa.21.9.3. PMID 21241645
- [Background] Carroll R, Meis M, Schulte M, Vormann M, Kiessling J, Meister H. Development of a German reading span test with dual task design for application in cognitive hearing research. Int J Audiol. 2015 Feb;54(2):136-41. doi: 10.3109/14992027.2014.952458. Epub 2014 Sep 8. PMID 25195607
- [Background] Zhong N, Jiang H, Wu J, Chen H, Lin S, Zhao Y, Du J, Ma X, Chen C, Gao C, Hashimoto K, Zhao M. Reliability and validity of the CogState battery Chinese language version in schizophrenia. PLoS One. 2013 Sep 2;8(9):e74258. doi: 10.1371/journal.pone.0074258. eCollection 2013. PMID 24023931
- [Background] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- See also: platform used for the mindfulness training — https://newlife330.hk/